CLINICAL TRIAL: NCT07131644
Title: A Randomized Controlled Trial Comparing Three Sirolimus Discontinuation Strategies in Patients With Kaposiform Hemangioendothelioma
Brief Title: Sirolimus Discontinuation Strategies in Kaposiform Hemangioendothelioma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi Ji, MD, PhD, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20250611
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Kaposiform Hemangioendothelioma
Keywords: Kaposiform Hemangioendothelioma; Sirolimus; Discontinuation Strategies
MeSH Terms: conditions — Kaposiform Hemangioendothelioma | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Direct discontinuation group (Placebo Comparator): Sirolimus was gradually tapered and discontinued over a 2-month period.
  Interventions: Drug: Sirolimus
- Low-dose treatment group (Experimental): Low-dose sirolimus treatment was administered for 6 months (with blood levels maintained at 2-5 ng/mL), followed by gradual tapering and discontinuation over 2 months.
  Interventions: Drug: Sirolimus
- Intermittent treatment group (Experimental): Sirolimus was administered using a 3-days-on/4-days-off weekly schedule for 6 months, followed by gradual tapering and discontinuation over 2 months.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — Comparison of different sirolimus discontinuation strategies.

SUMMARY:
Sirolimus has demonstrated efficacy in the treatment of kaposiform hemangioendothelioma (KHE); however, a high rate of rebound growth following discontinuation has been reported, highlighting the clinical importance of establishing an appropriate withdrawal regimen.

ELIGIBILITY:
Inclusion Criteria:

* KHE patients who have received sirolimus treatment and met the criteria for drug discontinuation.
* With evaluable clinical or imaging parameters to monitor disease activity or recurrence.
* Patients or their guardians are able to understand the study and provide written informed consent.
* Hematologic and hepatic/renal function meet the safety criteria for drug administration.

Exclusion Criteria:

* Patients who are unable to comply with the follow-up or treatment schedule, potentially affecting the integrity of study data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-13 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Rebound growth rate of KHE | 12 months
  The primary endpoint is the rebound growth rate of KHE during the follow-up period.

SECONDARY OUTCOMES:
Incidence of disease sequelae | 12 months
  Incidence of disease sequelae, assessed by the number of participants who develop clinically confirmed sequelae during the follow-up period, as determined through questionnaires and clinical plus imaging evaluations.
Incidence of adverse events throughout the study. | 12 months
  Incidence of adverse events during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ji, PhD, Principal Investigator — Sichuan University West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou J, Lan Y, Qiu T, Zhang Z, Gong X, Zhang X, Yang C, Zhou Z, Zhang Y, Yang M, Fu J, He C, Peng Q, Hu F, Xia C, Kong F, Chen S, Ji Y. Efficacy and safety of high-vs low-dose sirolimus in patients with kaposiform hemangioendothelioma: A randomized clinical trial. J Am Acad Dermatol. 2025 Jul;93(1):124-131. doi: 10.1016/j.jaad.2025.03.023. Epub 2025 Mar 17. PMID 40107509
- [Background] Zhou J, Li Y, Qiu T, Gong X, Yang K, Zhang X, Zhang Z, Lan Y, Hu F, Peng Q, Zhang Y, Kong F, Chen S, Ji Y. Long-term outcomes of sirolimus treatment for kaposiform hemangioendothelioma: Continuing successes and ongoing challenges. Int J Cancer. 2023 Aug 1;153(3):600-608. doi: 10.1002/ijc.34509. Epub 2023 Mar 22. PMID 36916140
- [Background] Ji Y, Chen S, Zhou J, Yang K, Zhang X, Xiang B, Qiu T, Gong X, Zhang Z, Lan Y, Hu F, Kong F, Qiu Q, Zhang Y. Sirolimus plus prednisolone vs sirolimus monotherapy for kaposiform hemangioendothelioma: a randomized clinical trial. Blood. 2022 Mar 17;139(11):1619-1630. doi: 10.1182/blood.2021014027. PMID 35030255
- [Background] Zhou J, Yang K, Dai S, Qiu T, Zhang X, Gong X, Chen S, Ji Y. Clinical features and management of kaposiform hemangioendothelioma and tufted angioma: Similarities and differences. J Am Acad Dermatol. 2022 Jul;87(1):172-174. doi: 10.1016/j.jaad.2021.07.012. Epub 2021 Jul 14. No abstract available. PMID 34273457
- [Background] Zhou J, Qiu T, Zhang Z, Lan Y, Huo R, Xiang B, Chen S, Qiu L, Xia C, Xu X, Li J, Ma Y, Yao W, Wang Z, Dong C, Qin Z, Tai M, Guo L, He X, Gu S, Li L, Hou F, Cai Y, Wang H, Wang J, Jiang X, Zheng J, Li K, Ji Y. Consensus statement for the diagnosis, treatment, and prognosis of kaposiform hemangioendothelioma. Int J Cancer. 2025 May 15;156(10):1986-1994. doi: 10.1002/ijc.35344. Epub 2025 Jan 20. PMID 39831682